CLINICAL TRIAL: NCT05795348
Title: ForceLoss: Part II - Osteoarthritic Patients. Development and Validation of Methods to Generate Personalised Models for the Differential Diagnosis of the Loss of Muscle Force
Brief Title: Personalised Modeling and Simulations for the Differential Diagnosis of Dynapenia: Study on Patients With Osteoarthritis
Acronym: ForceLoss II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ForceLoss II
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Dynapenia; Osteoarthritic patients; In Silico Medicine; Digital Twins; Maximal Voluntary Isometric Contraction; Musculoskeletal Modeling; Dynamometry; Electromyography; Superimposed Neuromuscular Electrical Stimulation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Knee Osteoarthritic Patients (Other): Patients candidate for knee arthroplasty; Age: 65-80 years; Body Mass Index: 18.5-30 kg/m²; ASA Classification: 1 or 2; Diagnosis of primary osteoarthritis at the knee; Suspect sarcopenia.
  Interventions: Diagnostic Test: Personalised Musculoskeletal Modeling

INTERVENTIONS:
Diagnostic Test: Personalised Musculoskeletal Modeling — Magnetic resonance images, electromyography and dynamometry data will be used to develop and inform personalised musculoskeletal models
  Other Names: Clinical measures (BIA, Hand-grip test); Clinical questionnaires (WOMAC, KSS)

SUMMARY:
The ForceLoss study aims to develop personalised modeling and simulation procedures to enable the differential diagnosis for the loss of muscle force, namely dynapenia. The primary causes of dynapenia can be identified in a diffuse or selective sarcopenia, a lack of activation (inhibition), or suboptimal motor control. Each of these causes requires different interventions, but a reliable differential diagnosis is currently impossible. While biomedical instruments and tools can provide valuable information, it is often left to the experience of the single clinican to integrate such information into a complete diagnostic picture. An accurate diagnosis for dynapenia is important for a number of pathologies, including neurological diseases, age-related frailty, diabetes, and orthopaedic conditions.

The hypothesis is that the use of mechanistic, subject-specific models (digital twins) to simulate a maximal isometric knee extension task, informed by experimental measures may be employed to conduct a robust differential diagnosis for dynapenia.

In this study, on patients candidate for knee arthroplasty, the investigators will expand (i) the experimental protocol previously developed and tested on healthy volunteers with a measure of involuntary muscle contraction (superimposed neuromuscular electrical stimulation, SNMES), a hand-grip test, measures of bio-impedance and clinical questionnaires, and (ii) the modeling and simulation framework to include one additional step (to check for muscle inhibition).

Medical imaging, electromyography (EMG) and dynamometry data will be collected and combined to inform a digital twin of each participant. Biomechanical computer simulations of a Maximal Voluntary Isometric Contraction (MVIC) task will then be performed. Comparing the models' estimates to in vivo dynamometry measurements and EMG data, the investigators will test one by one the three possible causes of dynapenia, and, through a process of hypothesis falsification will exclude those that do not explain the observed loss of muscle force.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Arthrosis at the knee (according to the American College of Rheumatology criteria), subjects elected for tota knee arthroplasty
* Body Mass Index between 18.5 and 30 kg/m2
* Health status (according to the American Society of Anesthesiology classification) equal to 1 or 2
* Suspected systemic sarcopenia due to aging or localized sarcopenia due to disuse

Exclusion Criteria:

* Neurological, rheumatic or tumoral diseases
* Inguinal or abdominal hernia
* Diabetes
* Severe Hypertension (Level 3)
* Severe Cardio-pulmonary insufficiency
* Diagnosis of Osteonecrosis in the lower limb joints
* Pathologies or physical conditions incompatible with the use of magnetic resonance imaging and electrostimulation (i.e., active and passive implanted biomedical devices, epilepsy, severe venous insufficiency in the lower limbs)
* Previous interventions or traumas to the joints of the lower limb

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Muscle volume | at baseline (Day 0)
  Full lower limb MRI data will be acquired with subjects in supine position. Individual muscle volumes (in cm3) will be segmented using commercial software and stored in anonymized form.
MVIC Torque | at baseline (Day 0)
  Dynamometry data will be acquired while participants perform a MVIC leg extension test. The maximum torque values (Nm) measured over three repetitions will be recorded. These correspond to the values observed in correspondence of the plateaux of force, developed over a sustained contraction.
Muscle Inhibition level | at baseline (Day 0)
  The difference between the maximal force exerted during the MVIC test (voluntary contraction) and that achieved when the muscles are electrically stimulated (involuntary contraction) will be computed.
Co-contraction index (CCI) | at baseline (Day 0)
  Experimental EMG data will be recorded from the major lower limb muscles involved in the knee extension, while participants perform a maximal voluntary isometric contraction on a dynamometer (i.e., MVIC test to quantify muscle strength).
  The co-contraction index, defined as the relative activation of agonist and antagonist muscles (for this task: quadriceps and hamstrings) in the act of kicking (MVIC test), will be computed according to Li et al (2020).

CONTACTS AND LOCATIONS:
Overall Officials: Marco Viceconti, Professor, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
We plan to share a database of experimental data representative of a population of patients elected for total knee arthroplasty. The dataset will include torques profiles and EMG data recorded during the MVIC test, the torque profiles recorded while delivering the electrical stimulation, and may include processed Magnetic Resonance Imaging data (segmentations of lower limb bones bones and muscles). All data will be irreversibly anonymized.
Time Frame: The (anonymized) dataset will be made available to the wider biomechanical community upon study completion
Access Criteria: Not yet defined

REFERENCES:
- [Background] Fernandez J, Zhang J, Heidlauf T, Sartori M, Besier T, Rohrle O, Lloyd D. Multiscale musculoskeletal modelling, data-model fusion and electromyography-informed modelling. Interface Focus. 2016 Apr 6;6(2):20150084. doi: 10.1098/rsfs.2015.0084. PMID 27051510
- [Background] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Background] Petterson SC, Barrance P, Buchanan T, Binder-Macleod S, Snyder-Mackler L. Mechanisms underlying quadriceps weakness in knee osteoarthritis. Med Sci Sports Exerc. 2008 Mar;40(3):422-7. doi: 10.1249/MSS.0b013e31815ef285. PMID 18379202
- [Background] Rice DA, McNair PJ. Quadriceps arthrogenic muscle inhibition: neural mechanisms and treatment perspectives. Semin Arthritis Rheum. 2010 Dec;40(3):250-66. doi: 10.1016/j.semarthrit.2009.10.001. Epub 2009 Dec 2. PMID 19954822
- [Background] Pons C, Borotikar B, Garetier M, Burdin V, Ben Salem D, Lempereur M, Brochard S. Quantifying skeletal muscle volume and shape in humans using MRI: A systematic review of validity and reliability. PLoS One. 2018 Nov 29;13(11):e0207847. doi: 10.1371/journal.pone.0207847. eCollection 2018. PMID 30496308
- [Background] Manini TM, Clark BC. Dynapenia and aging: an update. J Gerontol A Biol Sci Med Sci. 2012 Jan;67(1):28-40. doi: 10.1093/gerona/glr010. Epub 2011 Mar 28. PMID 21444359
- [Background] O'Brien TD, Reeves ND, Baltzopoulos V, Jones DA, Maganaris CN. The effects of agonist and antagonist muscle activation on the knee extension moment-angle relationship in adults and children. Eur J Appl Physiol. 2009 Aug;106(6):849-56. doi: 10.1007/s00421-009-1088-4. Epub 2009 May 27. PMID 19471955